CLINICAL TRIAL: NCT05867199
Title: Effects of Action Observation Therapy and Motor Imagery Administered During Immobilization Period After Surgical Fixation of Distal Radius
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CFL22/08
Record Dates: First submitted 2023-04-18; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Distal Radius Fracture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MI+AOT (Experimental): Subjects assigned to this group will be asked to perform Motor Imagery and Action Observation Training during immobilisation period after surgery. The training will be performed once a day, for three weeks. The duration of the training will last about 15 minutes.
  Interventions: Behavioral: Motor Imagery and Action Observation Training
- Control (No Intervention): Subjects assigned will be asked to follow standard care pathway during immobilisation period.

INTERVENTIONS:
Behavioral: Motor Imagery and Action Observation Training — The training consists of watching videos of actions performed with the hand. At the end of the video the subject is subsequently asked to imagine performing the action just seen
  Arms: MI+AOT

SUMMARY:
The goal of this trial is to verify the effectiveness of Motor Imagery and Action Observation Training in subjects undergoing surgery for distal radius fracture fixation. The main question it aims to answer is:

- can action observation and motor imagery training administered during immobilisation period improve functional outcome after distal radius fracture fixation? Participants will be asked to perform hand dexterity test and grip and pinch strength evaluation Subjects assigned to control group will follow standard care

ELIGIBILITY:
Inclusion Criteria:

* Right handed subjects
* Subjects after surgical distal radius fracture fixation

Exclusion Criteria:

* Concomitant fractures of upper limbs
* Pathological fractures
* Cognitive or psychiatric disorders
* Neurological or reumatici diseases

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Change of Purdue Pegboard Test score | After surgery (T0); 3 weeks after surgery (T1); 8 weeks after surgery (T2); 6 motnhs after surgery (T3)
  Change of Hand Dexterity test

SECONDARY OUTCOMES:
Change of Grip test | After surgery (T0); 3 weeks after surgery (T1); 8 weeks after surgery (T2); 6 motnhs after surgery (T3)
  Change in Grip strength evaluation with Jamar dynamometer
Change of Pinch test | After surgery (T0); 3 weeks after surgery (T1); 8 weeks after surgery (T2); 6 motnhs after surgery (T3)
  Change of Pinch strength evaluation
Change of Range of motion | After surgery (T0); 3 weeks after surgery (T1); 8 weeks after surgery (T2); 6 motnhs after surgery (T3)
  Change of Flexion, Extension, Ulnar deviation, Radial Deviation, Supination and Pronation measurement

OTHER OUTCOMES:
Change of Patient Rated Wrist Hand Evaluation | After surgery (T0); 3 weeks after surgery (T1); 8 weeks after surgery (T2); 6 motnhs after surgery (T3)
  Questionnaire about self reported rating of Hand and Wrist functionality

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided